CLINICAL TRIAL: NCT06452810
Title: A Clinical Trial to Evaluate the Effects of a Skin Balm on the Appearance of the Eye Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahajan (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20407
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Skin Health
Keywords: Eye Balm; Periorbital area; Dermatology

STUDY DESIGN:
Intervention Model Description: Study Type:
  Interventional (Clinical Trial)
  Estimated Enrollment:
  35 participants
  Allocation:
  Non-randomized
  Intervention Model:
  Single Group Assignment
  Masking:
  None (Open Label)
  Primary Purpose:
  Treatment
Masking Description: Masking:
  None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): All participants in this arm will receive the Sahajan Golden Glow Balm and will follow the same intervention protocol.
  Interventions: Dietary Supplement: Experimental: Sahajan Golden Glow Balm

INTERVENTIONS:
Dietary Supplement: Experimental: Sahajan Golden Glow Balm — Participants will apply the Sahajan Golden Glow Balm twice daily (morning and night) to the periorbital area following the specified instructions.

SUMMARY:
This virtual single-group clinical trial aims to evaluate the effects of the Sahajan Golden Glow Balm on the health and appearance of the skin in the periorbital area over a period of 6 weeks. Participants will apply the product twice daily and complete questionnaires at various intervals. Photos for expert skin grading will be taken at Baseline and Week 6.

DETAILED DESCRIPTION:
The study will investigate the impact of Sahajan Golden Glow Balm on skin health, particularly focusing on fine lines, wrinkles, dark circles, and dry eyes. It involves 35 female participants aged 35 and above, who will use the product for 6 weeks and complete periodic questionnaires and provide photos for dermatological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Concerns with the appearance of skin in the periorbital area
* Willing to maintain the same skincare routine for the study duration
* Must own a smartphone or digital camera for photos

Exclusion Criteria:

* Medical conditions affecting skin health
* Use of medications or products that could affect skin health
* Pregnancy or breastfeeding
* Participation in another clinical study

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Changes in the Health and Appearance of the Skin in the Periorbital Area | Baseline to Week 6
  The primary outcome measure will assess changes in the health and appearance of the skin in the periorbital area, evaluated via expert skin grading by a board-certified dermatologist.

SECONDARY OUTCOMES:
Changes in Participants' Perception of the Appearance of the Skin in the Periorbital Area | Baseline, Day 1, Week 2, Week 4, and Week 6
  The secondary outcome measure will evaluate changes in participants' perception of the appearance of their skin in the periorbital area, including the appearance of fine lines, wrinkles, dark circles, and dry skin, using participant-reported questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with study participants and published in open-access preprint servers following study completion and analysis.